CLINICAL TRIAL: NCT03120208
Title: Prevalence of Psychological Disorders After Immediate Postpartum Hemorrhage
Acronym: PSYCHE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHU-314; 2016-A00092-49 (Other: 2016-A00092-49)
Record Dates: First submitted 2017-04-07; First posted 2017-04-19 (Actual); Last update posted 2018-12-31 (Actual); Status verified 2018-12

CONDITIONS: Postpartum Hemorrhage; Postpartum Women; Postpartum Depression; Postpartum Stress; Postpartum Anxiety
Keywords: Postpartum psychological disorders; immediate postpartum hemorrhage.
MeSH Terms: conditions — Postpartum Hemorrhage; Depression, Postpartum | interventions — Psychiatric Status Rating Scales

STUDY DESIGN:
Masking Description: open
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- women in the nonexposed group without a hemorrhage (Experimental)
  Interventions: Behavioral: • The Edinburgh postnatal depression scale (EPDS), validated in French, with a discrimination threshold ≥ 11.; Behavioral: The GAD-7 with a discrimination threshold ≥10.; Behavioral: • Spielberger's State-Trait anxiety inventory, Form Y (validated in French), with a STAI (form Y-A) discrimination threshold ≥ 46; Behavioral: The IES-R, validated in French, with a discrimination threshold ≥ 30.
- women in the exposed group with a hemorrhage (Experimental)
  Interventions: Behavioral: • The Edinburgh postnatal depression scale (EPDS), validated in French, with a discrimination threshold ≥ 11.; Behavioral: The GAD-7 with a discrimination threshold ≥10.; Behavioral: • Spielberger's State-Trait anxiety inventory, Form Y (validated in French), with a STAI (form Y-A) discrimination threshold ≥ 46; Behavioral: The IES-R, validated in French, with a discrimination threshold ≥ 30.
- Partners (Experimental)
  Interventions: Behavioral: EPDS, MINI, STAI-A and B, IES-R and QEVA (experience)

INTERVENTIONS:
Behavioral: • The Edinburgh postnatal depression scale (EPDS), validated in French, with a discrimination threshold ≥ 11. — The Edinburgh postnatal depression scale (EPDS), validated in French, with a discrimination threshold ≥ 11.
  Arms: women in the exposed group with a hemorrhage; women in the nonexposed group without a hemorrhage
Behavioral: The GAD-7 with a discrimination threshold ≥10. — The GAD-7 with a discrimination threshold ≥10.
  Arms: women in the exposed group with a hemorrhage; women in the nonexposed group without a hemorrhage
Behavioral: • Spielberger's State-Trait anxiety inventory, Form Y (validated in French), with a STAI (form Y-A) discrimination threshold ≥ 46 — Spielberger's State-Trait anxiety inventory, Form Y (validated in French), with a STAI (form Y-A) discrimination threshold ≥ 46
  Arms: women in the exposed group with a hemorrhage; women in the nonexposed group without a hemorrhage
Behavioral: The IES-R, validated in French, with a discrimination threshold ≥ 30. — The IES-R, validated in French, with a discrimination threshold ≥ 30.
  Arms: women in the exposed group with a hemorrhage; women in the nonexposed group without a hemorrhage
Behavioral: EPDS, MINI, STAI-A and B, IES-R and QEVA (experience) — For the partners
  Arms: Partners

SUMMARY:
The objective of this cross-sectional study is to assess the prevalence of depression at 2 months, 6 months, and 1 year postpartum in women who had an immediate postpartum hemorrhage (immediate PPH defined as blood loss ≥ 500 mL within 24 hours of delivery). The potential serious consequences of PPH may lead to a greater number of psychological disorders in these women than in women without PPH.

DETAILED DESCRIPTION:
Study design: This repeated, cross-sectional, descriptive and etiological single-center study will take place within a cohort of women giving birth at the Clermont-Ferrand University Hospital Center (Psyche 1), and a cohort of their partners (psyche 2).

Principal endpoint: The prevalence of depression, measured by the Edinburgh postnatal depression scale (EPDS), validated in French, with a discrimination threshold ≥ 11.

Study plan and procedures:

Psyche 1:

For each woman with a PPH (exposed), 2 women without PPH (not exposed) will be included: the women who gave birth immediately before and immediate after her. If one of these 2 unexposed women eligible for the unexposed group also has a postpartum hemorrhage, another woman immediately just before or after the woman with PPH will be included. The PPH will be managed according to the national guidelines issued in December 2014.

The intervention will consist of 3 questionnaire surveys, at 2 months, 6 months, and 1 year postpartum.

Information and inclusion will take place in the immediate postpartum period at the Clermont-Ferrand University Hospital Center, France. An investigator (midwife or gynecologist-obstetrician in the maternity ward) will inform eligible women about the study, in the postpartum period. This investigator will provide them with a written information sheet and obtain their written consent. If the woman has already left the maternity ward, an investigator will contact her by mail or telephone, and she will receive the information sheet and consent form at her postnatal consultation in the department.

The cohort will complete each questionnaire at the same times in relation to their date of delivery (2 months, 6 months, and 12 months after). They will receive an email asking them to complete the questionnaires, including a participation number and an internet link to the self-administered questionnaires. This intervention is not usually performed for women who give birth at our hospital, whether or not they had a PPH. The procedures, other than the surveys, will be those provided habitually as usual care and will comply with good clinical practices and French regulations (1992 decree, French early discharge guideline from 2004). Should the questionnaire identify a woman in need of immediate psychological care, she will be contacted, referred to, and encouraged to consult a competent professional (psychologist, psychiatrist, child psychiatrist, etc.).

Psyche 2:

The cohort of partners will complete each questionnaire at the same times in relation to the date of delivery (2nd month and 6th month). The "source" documents will be the parturient's medical file (the part concerning both partners) and questionnaires, as the study involves a survey of the partners of women giving birth. The relevant covariables (confounding and prognostic factors) will also be collected from the women's medical files (emergency cesarean, vascular embolization, etc.). These covariables are already being collected as part of the Psyche 1 study.

Inclusion will take place in the immediate postpartum period. Accordingly, in the Psyche 1 study, for every woman with a PPH (exposed), 2 women without PPH (not exposed) are eligible (the woman who gave birth before and after the exposed woman). In this ancillary study, the partners, if eligible, of both the exposed and nonexposed women in the Psyche 1 study will be asked to participate.

The intervention will consist of 3 surveys by questionnaires: during the woman's hospitalization during the immediate postpartum period, at 2 months, and at 6 months after the delivery.

The partners of the women who had an immediate postpartum hemorrhage (PPH) will be compared to the partners of the women who did not.

Data collection:

The source documents will be the medical file and the questionnaires. Clinicians will make the data extraction from the medical files, including the relevant covariables: confounding factors, prognostic factors (e.g., history of depression, anxiolytic treatment before delivery, psychological or psychiatric care before and delivery and after delivery, etc.).

Quality assurance plan:

* The Investigator undertakes to conduct this study in compliance with Good Clinical Practices and French public health law [Act n°2004-806 dated 9 August 2004 concerning biomedical research, its implementing decree n° 2006-477 dated 26/04/2006, which modifies the portion of the Public Health Code (specifically, Part 1, Book 1, Title II, Section 1) concerning biomedical research, as well as the decrees in force]. The investigator also undertakes to conduct this research in accordance with Declaration of Helsinki of the World Medical Association (Tokyo 2004, as revised).
* The investigators guarantee the authenticity of the data collected in this study and accept the legal provisions authorizing the study sponsor to set up quality control procedures. During quality control inspections, the following items will be checked:

  * Informed consent.
  * Compliance with the research protocol and the procedures defined there.
  * Assurance of the quality of the data collected in the electronic CRF: accuracy, missing data, consistency of the data with the source documents (such as paper and electronic medical files and questionnaires completed by the midwives).

Reporting for adverse events:

In compliance with decree n° 2006-477 dated 26/04/2006, which modifies the portion of the Public Health Code (specifically, Part 1, Book 1, Title II, Section 1) concerning biomedical research, as well as the decrees in force, any suspected unexpected serious adverse effect will be reported by the Sponsor to the competent, authority at the CPP, as soon as the Sponsor is aware of it and at the latest 7 days after the event.

Sample size assessment:

Psyche 1: For a power of 90%, with a two-sided alpha of 5%, with 2 unexposed subjects for 1 exposed and according to the Australian study by JF Thompson et al. (2011) who found a depression rate of 10% in unexposed and 16% in exposed women at 4 months postpartum, this study requires:

* 1028 women in the unexposed group, with no hemorrhage
* and 514 women in exposed group with a hemorrhage

A total of 1542 women must therefore be included.

Statistical analysis plan:

There will be 3 samples for analysis:

* Respondents to the survey at 2 months
* Respondents to the survey at 6 months
* Respondents to the survey at 12 months (not for partners)

The participation and refusal rates will be calculated at each survey point, together with the prevalence of the psychological states studied. Some women will be lost to follow-up at the M6 and M12 surveys. These women will be included in the crude descriptive analyses, and population lost to follow-up will be compared with the study population to look for possible differences in the principal characteristics studied. We plan to perform an interim analysis to assess the need to adjust the study calendar. This interim analysis will be performed after half of the planned subjects have been included.

Statistical techniques:

The statistical methods used for the crude analyses will be a descriptive analysis of the sample with a comparison of the exposed and unexposed groups, where we describe the characteristics of the groups included in the study.

The Chi 2 test (or Fisher's exact test when appropriate) will be used to compare the qualitative variables and Student's t test (or a Mann-Whitney test) for the quantitative variables.

Prevalence rates and their 95% confidence intervals will be calculated for depression at 2 months, 6 months, and 1 year.

A multivariate analysis (logistic regression) will be conducted to take into account confounding factors (smoking, cannabis, etc.) as well as clinically relevant prognostic factors (history of depression, use of anxiolytic or antidepressant agents, etc.) for depression at each survey interval (at 2 months, 6 months, and 1 year). The results will be expressed as adjusted odds ratios (aOR).

At the end of the study, another multivariate analysis (generalized linear mixed model) will be performed to study the trends in the prevalence of depression over the 3 study periods.

Plan for missing data

The missing data will be treated as missing and excluded from the analyses.

ELIGIBILITY:
For the women:

Inclusion criteria:

* women who gave birth at a term ≥ 22 weeks' gestation or, if the term is unknown, to a fetus with a birth weight ≥ 500 g),
* regardless of the type of delivery (vaginal or cesarean),
* regardless of parity or fetal presentation,
* and regardless of type of pregnancy (singleton or multiple).
* and affiliated with French CNAMTS (salaried worker) health insurance.

Exclusion criteria:

Women who are:

* minors,
* who do not understand French,
* who refuse to participate (did not sign consent),
* and who did not give birth at the Clermont-Ferrand University Hospital Center maternity unit and were secondarily transferred there postpartum.

For the partners:

Inclusion criteria:

* Partner of a woman who gave birth at a term ≥ 22 weeks of gestation or, if the term is unknown, to a fetus with a birth weight ≥ 500 g),
* Regardless of the type of delivery (vaginal or cesarean),
* Regardless of parity and fetal presentation,
* And regardless of type of pregnancy (singleton or multiple),
* And both partners are affiliated with French CNAMTS (salaried worker) health insurance.

Exclusion criteria:

* Partner of a woman who gave birth at a term < 22 weeks of gestation or, if the term is unknown, to a fetus with a birth weight < 500 g),
* Partner who does not understand French,
* Who refuses to participate (does not sign consent),
* Partner who is a minor,
* Protected adult,
* Partner not present at the maternity ward (woman is divorced, separated, has no partner, or the partner is abroad or in prison or died during pregnancy),
* And partners of women who gave birth outside the UHC and was transferred to it only secondarily in the postpartum period.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1968 (Estimated)
Dates: Start 2017-04-27 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
prevalence of depression | at 12 months after delivery.
  the prevalence of depression, measured by the Edinburgh postnatal depression scale (EPDS), validated in French, with a discrimination threshold ≥ 11

SECONDARY OUTCOMES:
prevalence of depression among women with PPH between 500-1000 mL compared with those with severe PPH (≥ 1000 mL) | at 2 months, 6 months, and 12 months after delivery.
  prevalence of depression among women with PPH between 500-1000 mL
The prevalence of depression among women with a PPH requiring a so-called second-order medical intervention (transfusion, vascular embolization, etc.) compared with women who had a PPH without such a second-order intervention | at 2 months, 6 months, and 12 months after delivery
  The prevalence of depression among women with a PPH requiring a so-called second-order medical intervention (transfusion, vascular embolization, etc.) compared with women who had a PPH without such a second-order intervention
severity of depression among women with PPH between 500-1000 mL compared with those with severe PPH (≥ 1000 mL) | at 2 months, 6 months, and 12 months after delivery
  severity of depression among women with PPH between 500-1000 mL compared with those with severe PPH (≥ 1000 mL)
severity of depression among women with a PPH requiring a so-called second-order medical intervention (transfusion, vascular embolization, etc.) compared with women who had a PPH without such a second-order intervention | at 2 months, 6 months, and 12 months after delivery
  severity of depression among women with a PPH requiring a so-called second-order medical intervention (transfusion, vascular embolization, etc.) compared with women who had a PPH without such a second-order intervention
prevalence of anxiety and post-traumatic stress among women after an immediate PPH | at 2 months, 6 months, and 12 months after delivery
  prevalence of anxiety and post-traumatic stress among women after an immediate PPH
prevalence of anxiety and post-traumatic stress among women with PPH between 500-1000 mL compared with those with severe PPH (≥ 1000 mL) | at 2 months, 6 months, and 12 months after delivery
  prevalence of anxiety and post-traumatic stress among women with PPH between 500-1000 mL compared with those with severe PPH (≥ 1000 mL)
prevalence of anxiety and post-traumatic stress among women with a PPH requiring a so-called second-order medical intervention (transfusion, vascular embolization, etc.) compared with women who had a PPH without such a second-order intervention | at 2 months, 6 months, and 12 months after delivery
  prevalence of anxiety and post-traumatic stress among women with a PPH requiring a so-called second-order medical intervention (transfusion, vascular embolization, etc.) compared with women who had a PPH without such a second-order intervention
severity of anxiety and post-traumatic stress among women with PPH between 500-1000 mL compared with those with severe PPH (≥ 1000 mL) | at 2 months, 6 months, and 12 months after delivery
  severity of anxiety and post-traumatic stress among women with PPH between 500-1000 mL compared with those with severe PPH (≥ 1000 mL)
severity of anxiety and post-traumatic stress among women with a PPH requiring a so-called second-order medical intervention (transfusion, vascular embolization, etc.) compared with women who had a PPH without such a second-order intervention | at 2 months, 6 months, and 12 months after delivery
  severity of anxiety and post-traumatic stress among women with a PPH requiring a so-called second-order medical intervention (transfusion, vascular embolization, etc.) compared with women who had a PPH without such a second-order intervention
prevalence of depression, post-traumatic stress, and anxiety, the experience of delivery, in partners of women with an immediate postpartum hemorrhage (< 24 hours) | at 2 months and 6 months after the woman gave birth.

CONTACTS AND LOCATIONS:
Overall Officials: Marine PRANAL JULIEN, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Pranal M, Legrand A, de Chazeron I, Llorca PM, Vendittelli F. Prevalence of maternal psychological disorders after immediate postpartum haemorrhage: a repeated cross-sectional study - the PSYCHE* study protoco. BMJ Open. 2019 Sep 4;9(9):e027390. doi: 10.1136/bmjopen-2018-027390. PMID 31488469